CLINICAL TRIAL: NCT02777281
Title: Safe and Effective Shoulder Exercise Training in Manual Wheelchair Users With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1405M50661
Record Dates: First submitted 2014-05-14; First posted 2016-05-19 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Shoulder Pain; Spinal Cord Injury
Keywords: Shoulder Pain; Wheelchair; Spinal Cord injury
MeSH Terms: conditions — Shoulder Pain; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shoulder pain and SCI (Other): Manual wheelchair users with SCI
  Interventions: Behavioral: Shoulder pain and SCI
- Shoulder pain and able bodies (Other): No SCI or wheelchair use but presence of shoulder pain
  Interventions: Behavioral: Shoulder pain and able bodies

INTERVENTIONS:
Behavioral: Shoulder pain and SCI — Shoulder pain and SCI
  Arms: Shoulder pain and SCI
Behavioral: Shoulder pain and able bodies
  Arms: Shoulder pain and able bodies

SUMMARY:
This study will compare two exercise programs in an interventional study for manual wheelchair users with spinal cord injury and shoulder pain. Subjects without spinal cord injury will also be enrolled to compare exercise approaches.

DETAILED DESCRIPTION:
The investigators hypothesis is that the biomechanically based exercise program will demonstrate greater muscle activation of targeted muscles, and reduced compression risk to the rotator cuff tendons.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with paraplegia at least 1 year post SCI. Prior to this time patients are still adjusting to independent function with manual wheelchairs as their primary means of mobility. This criteria ensures the subjects have had sufficient exposure to the functional demands associated with their condition.
2. Age 21 to 60 years old; below age 21, particularly in males, the humeral growth plate may not have fully closed. Including subjects above this age ensures skeletal maturity. After age 60, even in able-bodied individuals, substantial degenerative changes can begin to occur in the shoulder joint.
3. Use of a manual wheelchair as the primary means of mobility (> 50% time). This is the population with most risk of development of shoulder pain and associated secondary complications.
4. A history of unilateral or bilateral shoulder pain that interferes with at least one functional task. Symptoms localized to the proximal anterior, lateral, or posterior glenohumeral (shoulder joint) region are required. Rotator cuff tendinopathy and "impingement" syndromes involve localized pain in this region. More diffuse symptoms are consistent with combined shoulder/neck syndromes or radiating pain from cervical spine pathology.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Reproduction of shoulder pain, pain radiating down the upper extremity, numbness or tingling in the upper extremity, or other upper extremity symptoms during a cervical screening examination or thoracic outlet testing. This result would be indicative of primary cervical or thoracic outlet pathology.
3. Shoulder pain of traumatic origin. Cumulative trauma disorders are of primary interest and most amenable to the proposed exercise interventions.
4. History of shoulder surgery or dislocation.
5. Recent history of fracture (within 1 year), hospitalization (within the past month), or cortisone injection to the shoulder (within 4 months). These conditions may interfere with safe or effective completion of the exercise intervention.
6. A diagnosis or imaging findings of rheumatoid arthritis, end stage osteoarthritis, full thickness rotator cuff tear, adhesive capsulitis, or complex regional pain syndrome. These subjects may have joint disease progression that is severe, or not appropriately treated with a stretching and strengthening intervention.
7. Diagnosed major depression, alcohol or substance abuse, or other serious medical conditions. These conditions may prevent subjects from regularly completing the exercise intervention

All criteria apply to both groups excepting manual wheelchair use and SCI criteria not applicable to the able bodied subject group.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Muscle activity | baseline
  Muscle activity during exercises is measured as a change in EMG
Rotator cuff compression risk | baseline
  Motion and position data of the upper arm relative to the shoulder blade measured in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Ludewig, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States